CLINICAL TRIAL: NCT03171818
Title: Darbepoetin for Ischemic Neonatal Stroke to Augment Regeneration
Acronym: DINOSAUR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Collaborators: Alberta Children's Hospital (Other); The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, dr. M.J.N.L. Benders, Principal Investigator UMC Utrecht, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL53975.041.16
Record Dates: First submitted 2017-05-24; First posted 2017-05-31 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: PAIS; Neonatal Stroke; Perinatal Stroke
MeSH Terms: interventions — Darbepoetin alfa; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: An international multicenter, randomized placebo controlled intervention study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This will be a double-blinded study, meaning that both the patient (and his/her parents) and the health care providers, including neonatologist, pediatrician, nurses, physiotherapists, etc, are not allowed to know what treatment the patient has been given. Those that collect outcome parameters, such as MRI data and neurodevelopmental outcome, are also unaware of treatment allocation, meaning that blinding will be maintained during the full study-period of 18 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Darbepoetin (Experimental): Darbepoetin alfa (Aranesp, Amgen)
  Interventions: Drug: Darbepoetin Alfa
- Placebo (Placebo Comparator): Saline
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Darbepoetin Alfa — Darbepoetin alfa (Aranesp, Amgen) 2 doses of 10 microgram/kg i.v.
  Other Names: Aranesp
  Arms: Darbepoetin
Drug: Saline — The placebo will consist of saline, containing 9.0 g of salt per liter (0.90%) i.v.
  Other Names: Sodium Chloride
  Arms: Placebo

SUMMARY:
The aim of the study is to perform a randomized double-blind placebo controlled prospective study in newborn infants with MRI confirmed Middle Cerebral Artery (MCA) Perinatal Arterial Ischemic Stroke (PAIS) with darbepoetin. It will be investigated whether intravenous administered darbepoetin can induce the formation of neuronal tissue and restore brain function in neonates who suffered from PAIS compared to placebo treated controls. The ultimate goal of this study is therefore to develop a therapy using erythropoiesis-stimulating agents (ESA) such as darbepoetin to reduce or even prevent lifelong consequences of PAIS-related brain injury in this group of term newborns.

ELIGIBILITY:
Inclusion Criteria:

* Newborns ≥ 36+0 weeks of gestation, both male and female
* MRI confirmed diagnosis of acute PAIS, in the MCA region with involvement of the cortical spinal tract (e.g. Posterior Limb of Internal Capsule [PLIC] or peduncles) within one week after birth
* Written informed consent from custodial parent(s)

Exclusion Criteria:

* Moderate -severe Hypoxic-Ischemic Encephalopathy (HIE) with or without hypothermia therapy
* Any proven or suspected major congenital anomaly, chromosomal disorder, metabolic disorder;
* Presence of a serious infection of the central nervous system;
* No realistic prospect of survival, (e.g. severe brain injury), at the discretion of the attending physician.
* Infant for whom withdrawal of supportive care is being considered.

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in stroke tissue loss | 6-8 weeks of age
  The primary objective is to determine whether there is a difference in the degree in stroke tissue loss between darbepoetin and placebo treatment, which will be measured by the change in lesion size between the time of onset of the insult and 6-8 weeks of age. The primary endpoint will be estimated using advanced volumetric magnetic resonance (MRI) techniques, performed within one week after clinical presentation and at 6-8 weeks of age.

SECONDARY OUTCOMES:
Reorganization of corticospinal connectivity | 6-8 weeks of age
  To assess whether there are differences between darbepoetin and placebo treatment in Diffusion Tensor Imaging (DTI) parameters of selected regions of interest. DTI-MRI techniques are performed at 6-8 weeks of age.
Neurodevelopment | 18 months of age
  To assess cognitive and motor development at 18 months of age using the Bayley Scales of Infants and Toddler Development (BSITD)-III scores compare them between groups (darbepoetin vs placebo).
Neurological assessment | 18 months of age
  To assess neurological deficit and function using the Pediatric Stroke Outcome Measure (PSOM) and compare this score between groups (darbepoetin vs placebo). The PSOM is performed at 18 months of age.
Development of Cerebral Palsy | 18 months of age
  Development of Unilateral Spastic Cerebral Palsy (USCP) using the Gross Motor Function Classification system (GMFCS) and compare this between groups (darbepoetin vs placebo).

CONTACTS AND LOCATIONS:
Overall Officials: Manon Benders, MD PhD, Principal Investigator — UMC Utrecht
Locations (1):
- Wilhelmina Childrens Hostpital/University Medical Center Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benders MJ, van der Aa NE, Roks M, van Straaten HL, Isgum I, Viergever MA, Groenendaal F, de Vries LS, van Bel F. Feasibility and safety of erythropoietin for neuroprotection after perinatal arterial ischemic stroke. J Pediatr. 2014 Mar;164(3):481-6.e1-2. doi: 10.1016/j.jpeds.2013.10.084. Epub 2013 Dec 8. PMID 24321539